CLINICAL TRIAL: NCT02989727
Title: Melancholic Symptoms in Bipolar Depression and Responsiveness to Lamotrigine: Results From an 8-week, Multicenter, Double-blind, Placebo-controlled Trial
Brief Title: Melancholic Symptoms in Bipolar Depression and Responsiveness to Lamotrigine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Evyn Peters, Resident, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSK-SCA100223
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Depression; Bipolar Disorder; Bipolar Depression; Melancholia; Lamotrigine
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lamotrigine - melancholic depression (Experimental): Participants with melancholic depression who were randomly assigned to receive lamotrigine tablets escalated to a target dose of 200mg/day.
  Interventions: Drug: Lamotrigine
- Placebo - melancholic depression (Placebo Comparator): Participants with melancholic depression who were randomly assigned to receive a placebo comparator.
  Interventions: Drug: Placebos
- Lamotrigine - nonmelancholic depression (Experimental): Participants not meeting DSM-IV-TR diagnostic criteria for melancholic depression who were randomly assigned to receive lamotrigine tablets escalated to a target dose of 200mg/day.
  Interventions: Drug: Lamotrigine
- Placebo - nonmelancholic depression (Placebo Comparator): Participants not meeting DSM-IV-TR diagnostic criteria for melancholic depression who were randomly assigned to receive a placebo comparator.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine tablets at dosages of 25mg/day for Week 1 and Week 2, 50mg/day for Week 3 and Week 4, 100mg/day for Week 5, and 200mg/day for Week 6, Week 7, and Week 8.
  Other Names: Lamictal
  Arms: Lamotrigine - melancholic depression; Lamotrigine - nonmelancholic depression
Drug: Placebos — Placebo tablets
  Other Names: Placebo
  Arms: Placebo - melancholic depression; Placebo - nonmelancholic depression

SUMMARY:
The purpose of this study is to determine if patients with melancholic bipolar II depression are more responsive to lamotrigine than patients with non-melancholic bipolar II depression. To do this, the investigators will re-analyze a previous clinical trial that evaluated lamotrigine as a treatment for bipolar II depression (GSK-SCA100223; NCT00274677).

DETAILED DESCRIPTION:
Patients suffering from depression with melancholic symptoms (i.e., anhedonia, flat affect, diurnal mood variation, terminal insomnia, psychomotor disturbances, decreased weight/appetite, and excessive guilt) respond better to certain antidepressants. Melancholic symptoms also occur in bipolar depression, although they have received less research. Lamotrigine has been shown to alter some of the biological processes that are known to occur in melancholic depression. The purpose of this study is to determine if patients with melancholic bipolar II depression are more responsive to lamotrigine than patients with non-melancholic bipolar II depression.

This study will re-analyze data from a previous 8-week, randomized, placebo-controlled trial that evaluated lamotrigine as a treatment for bipolar II depression (GSK-SCA100223; NCT00274677). The original study data was made available by GlaxoSmithKline as part of an initiative to make clinical trials data available for research use. Access was applied for via https://www.clinicalstudydatarequest.com.

The analysis strategy will be comparable to the original study, although the investigators will first classify participants as suffering from either melancholic or non-melancholic depression. The diagnosis of melancholic depression was established according to baseline responses to the Hamilton Depression Rating Scale (HAMD-17) and the Montgomery-Åsberg Depression Rating Scale (MADRS), according to the DSM-IV-TR diagnostic criteria. HAMD-17 and MADRS change scores will be compared between the treatment and placebo groups using Analysis of Variance (ANOVA). Both ANOVA models will include a test for an interaction between treatment group (lamotrigine vs. placebo) and melancholic depression (melancholic depression vs. non-melancholic depression). To handle missing data, each ANOVA model will be computed with only complete-case data first and subsequently using inverse probability weights that account for the probability of drop out. Inverse probability weights will be created based on covariates that predict missing responses. HAMD-17 and MADRS response rates between the treatment and placebo groups will be evaluated with a Cox proportional hazard regression analysis. There will be two separate analyses, one including participants with melancholic depression, and one including participants with non-melancholic depression. Statistical models will also adjust for baseline depression severity, if participants with melancholic depression are found to have more severe depressive symptoms at baseline.

Given the delay between antidepressant initiation and response, trial-and-error prescribing is an inevitably lengthy process. The investigators hope the results of this study will enable more timely and effective treatment for patients with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written and informed consent.
2. Diagnosis of Bipolar II Disorder and currently depressed for minimum of the last 8 weeks, with a HAMD-17 score of at least 18 with scores of 3 or more on Items 1 or 7.
3. For females, be of non-childbearing potential, or of childbearing potential with a negative pregnancy test at screening and agrees to one of (a) abstinence from sex two weeks prior and five days after drug continuation/discontinuation, (b) personal or partner sterilization, (c) one method of hormonal contraception, or (d) two barrier methods of contraception.
4. Acceptable results (within two times the normal limit) on laboratory screening tests (e.g., thyroid function).

Exclusion Criteria:

1. Active suicidality.
2. History of non-response to antidepressant treatment, or any previous treatment with lamotrigine.
3. History of substance dependence in the past year, or abuse within the 4 weeks prior to study entry.
4. Rapid cycling bipolar disorder.
5. Receiving additional psychoactive medication (not including lorazepam for agitation), or has started a new course of psychotherapy within the last month.
6. Received treatment for an anxiety or eating disorder within the last 12 months.
7. Investigational drug use within the last month.
8. History of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-11; Primary Completion 2005-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudy C Bowen, FRCPC, Study Director — University of Saskatchewan
Locations (1):
- Department of Psychiatry, Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for the study (GSK-SCA100223; NCT00274677) is available through www.clinicalstudydatarequest.com.

REFERENCES:
- See also: The ClinicalTrials.gov posting for the original study (GSK-SCA100223; NCT00274677) from which data for the present study was obtained. — https://clinicaltrials.gov/ct2/show/record/NCT00274677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study only analyzed data from treatment completers in the original study, NCT00274677. The original study enrolled 221 participants, with 150 completing the trial.
Period: Overall Study
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Started (We only analyzed data from treatment completers (n=150) in the original study (n=221), NCT00274677.) | 46 | 44 | 30 | 30
Completed | 46 | 44 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression | Total
Number analyzed (Participants) | 46 | 44 | 30 | 30 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.5) | 37.8 (10.9) | 41.2 (10.6) | 35.8 (11.2) | 38.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 19 | 17 | 99
  Male | 15 | 12 | 11 | 13 | 51

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Change Scores
Description: Scale scores range from 0 to 60. This outcome is a change score calculated by subtracting Baseline from Week 8 scores.
  Lower scores indicate greater improvement of depressive symptoms.
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
score on a scale | -15.7 (10.8) | -13.8 (11.6) | -16.0 (10.5) | -15.5 (9.93)
Statistical Analysis 1: Comparison: Lamotrigine - Melancholic Depression vs Placebo - Melancholic Depression vs Lamotrigine - Nonmelancholic Depression vs Placebo - Nonmelancholic Depression; Weighted ANOVA models were used to compare change scores between lamotrigine and placebo groups while testing for interactions by melancholic status. The estimate and test reported is for the the interaction between treatment condition and melancholic status; Test type: Superiority; p = .59, ANOVA; ANOVA estimate = 1.88, Standard Error of Mean 3.51

2. Primary Outcome: Hamilton Depression Rating Scale (HAMD-17) Change Scores
Description: Scale scores range from 0 to 52. This outcome is a change score calculated by subtracting Baseline from Week 8 scores.
  Lower scores indicate greater improvement of depressive symptoms.
Time Frame: Eight weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
score on a scale | -13.5 (7.92) | -10.9 (9.52) | -13.0 (7.59) | -10.6 (6.55)
Statistical Analysis 1: Comparison: Lamotrigine - Melancholic Depression vs Placebo - Melancholic Depression vs Lamotrigine - Nonmelancholic Depression vs Placebo - Nonmelancholic Depression; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .84, ANOVA; ANOVA estimate = 0.5, Standard Error of Mean 2.56

3. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Eight weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 28 | 22 | 20 | 16
Statistical Analysis 1: Comparison: Lamotrigine - Melancholic Depression vs Placebo - Melancholic Depression; Weighted Cox regression with treatment condition (lamotrigine vs. placebo) predicting treatment response. Response is defined as a score reduction of at least 50% from baseline. The outcome variable is binary coded with "1" being a response at anytime point and "0" indicating no response; Test type: Superiority; p = .08, Regression, Cox; Cox Proportional Hazard = 1.2, Standard Error of Mean .10
Statistical Analysis 2: Comparison: Lamotrigine - Nonmelancholic Depression vs Placebo - Nonmelancholic Depression; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .53, Regression, Cox; Cox Proportional Hazard = 1.08, Standard Error of Mean .12

4. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Seven weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 27 | 21 | 20 | 20

5. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 28 | 19 | 15 | 13

6. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Five weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 25 | 19 | 12 | 9

7. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 14 | 16 | 9 | 8

8. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 11 | 10 | 8 | 8

9. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Two weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 6 | 6 | 3 | 4

10. Primary Outcome: Number of Participants With 50% Reduction in the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Scale scores range from 0 to 60. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 5 | 3 | 2 | 2

11. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Eight weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 25 | 22 | 20 | 14
Statistical Analysis 1: Comparison: Lamotrigine - Melancholic Depression vs Placebo - Melancholic Depression; Weighted Cox regression with treatment condition (lamotrigine vs. placebo) predicting treatment response. Response is defined as a score reduction of at least 50% from baseline. The outcome variable is binary coded with "1" being a response at any time point and "0" indicating no response; Test type: Superiority; p = .02, Regression, Cox; Cox Proportional Hazard = 1.27, Standard Error of Mean .11
Statistical Analysis 2: Comparison: Lamotrigine - Nonmelancholic Depression vs Placebo - Nonmelancholic Depression; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = .73, Regression, Cox; Cox Proportional Hazard = 1.05, Standard Error of Mean .13

12. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Seven weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 28 | 19 | 15 | 18

13. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Six weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 29 | 17 | 14 | 11

14. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Five weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 22 | 19 | 10 | 9

15. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Four weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 16 | 13 | 9 | 11

16. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 11 | 9 | 8 | 7

17. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: Two weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 7 | 6 | 5 | 4

18. Primary Outcome: Number of Participants With 50% Reduction in the Hamilton Depression Rating Scale (HAMD-17)
Description: Scale scores range from 0 to 52. A response is defined as a score reduction from baseline of at least 50%.
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine - Melancholic Depression | Placebo - Melancholic Depression | Lamotrigine - Nonmelancholic Depression | Placebo - Nonmelancholic Depression
Number analyzed (Participants) | 46 | 44 | 30 | 30
Participants | 3 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: 8 weeks.
Description: We have combined the two lamotrigine arms (melancholic and nonmelancholic) into one group, and also the two placebo arms (melancholic and nonmelancholic) into one group. We did not analyze safety data by melancholic status, so we are only able to report the original safety results (which was stratified by treatment condition but not melancholic status).
Groups:
- Lamotrigine; Placebo: The data is from 109 participant that were randomized in the original trial.
Arm/Group | Lamotrigine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/109 | 5/109
Other Adverse Events (participants affected / at risk) | 88/109 | 85/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamotrigine (N=109) | Placebo (N=109)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=109) | Placebo (N=109)
Headache (Nervous system disorders) | 30 | 39
Dry mouth (General disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 9 | 7
Nasopharyngitis (General disorders) | 0 | 9
Nausea (Gastrointestinal disorders) | 8 | 15
Dizziness (General disorders) | 7 | 8
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Sedation (General disorders) | 6 | 2
Somnolence (General disorders) | 6 | 5
Fatigue (General disorders) | 3 | 7
Vomiting (Gastrointestinal disorders) | 2 | 6

LIMITATIONS AND CAVEATS:
1. Short duration of trial in context of slow dosing regime
2. Inability to assess other definitions of melancholia
3. Sample of only bipolar II depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No